CLINICAL TRIAL: NCT04651075
Title: Effects On Physıological Parameters And Anxiety Of Related Musıc And Informatıon Training Before Coronary Angiography
Brief Title: Music Listenıng And Training Before Coronary Angıography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIBU-HSF-AYN-01
Record Dates: First submitted 2020-06-26; First posted 2020-12-03 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease; Anxiety; Music; Education
Keywords: Coronary Angiography; Teaching; Music theraphy; Anxiety; Nursing care
MeSH Terms: conditions — Coronary Artery Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: There are 3 groups as intervention and control
Who Masked: Participant
Masking Description: the participant did not know which group he was in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- music theraphy (Experimental): One of the 4 music genres (Turkish Folk, Classical, Turkish Art and Sufi Music), which was determined by the researcher by scanning the literature 30 minutes before the CAG procedure, and the expert opinion was taken to the participants in this group was played with a 5-minute headset. The musical genres were arranged in instrumental, nonverbal, 70 decibels in terms of rhythm and duration and played according to the individual's choice.
  Interventions: Other: music listening
- information education (Experimental): Participants in this group were trained to inform them about CAG in visual, audio and written form. Information training was provided by the researcher 30 minutes before the CAG procedure after the outpatient clinic controls of the patient. Information education prepared by the researcher by scanning the literature and getting expert opinion; It includes 7 minutes of video explanation about the CAG process, discussion after video watching, question and answer, and the delivery of a training book prepared in written form.
  Interventions: Other: individual training
- nursing care (No Intervention): Individuals in this group received routine nursing care and no intervention was made by the researcher. In routine nursing care for individuals who will receive CAG procedure in the clinic; Preparation for the CAG procedure, which involves opening the vascular access and dressing the surgical gown, is included in the pre-and post-procedure routine once and more frequently when there are deviations from normal, and if the patient asks questions about the procedure, measurement of blood pressure, heart rate and oxygen saturation.

INTERVENTIONS:
Other: music listening — The music selected by the participants was played to the music listening group.
  Arms: music theraphy
Other: individual training — Individual training group was trained on coronary angiography.
  Arms: information education

SUMMARY:
The aim of this study was to investigate the effects of education and music listening on the anxiety and physiological parameters experienced by individuals undergoing elective coronary angiography.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of education and music listening on the anxiety and physiological parameters experienced by individuals undergoing elective coronary angiography.

The population of the study consisted of individuals undergoing elective coronary angiography in the Cardiology Department of Abant İzzet Baysal University İzzet Baysal Training and Research Hospital. The study was conducted in a randomized controlled manner with three groups: 34 individuals in music listening group (M1), 34 individuals in information training group (M2) and 34 subjects in control group. In order to collect data, CAG (Coronary angiography) Procedure Training Form, Patient Identification Form, Physiological Parameters Form and Visual Analogue Scale and Spielberg State and Trait Anxiety Scale were used. Data were collected by face to face interview technique. Descriptive statistics, Independet Simple test, Paired sample t test, Kruskall Wallis, Mann Whitney U test and Wilcoxon signed rank test were used in the analysis of the data and the significance level was accepted as p <0.05.

ELIGIBILITY:
Inclusion Criteria:

Applying femoral CAG electively,

* The first time CAG will be held,
* Performing the CAG procedure for diagnostic purposes,
* Not trained on the CAG process,
* Volunteering to participate in the study,
* No problem in verbal communication,
* No hearing loss,
* Being able to read and write,
* Has not been diagnosed with psychiatric illness,
* Being conscious,
* Being 18 or older.

Exclusion Criteria:

Radial application of CAG,

* Previously performing coronary angiography,
* Performing the CAG procedure for therapeutic purposes (stent, balloon, etc.),
* Having received training on the KAG process,
* Does not want to participate in the study
* Problems in verbal communication,
* Hearing loss,
* Psychiatric illness is found.
* Consciousness is closed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
means of subjective anxiety scores | up to 45 minutes
  Spielberg State- Trait Anxiety Scale. The total score between 0-19 obtained from the state anxiety scale shows that there is no anxiety, the total score between 20-39 indicates mild, the average score between 40-59 indicates moderate, and the total score between 60-79 indicates severe anxiety, and over 60 points are needed for professional help. The scores obtained from the trait anxiety scale vary between 20 and 80. A high score means a high and a low level means anxiety.

SECONDARY OUTCOMES:
means of subjective pain scores | up to 45 minutes
  visual analog scale. It consists of a straight line with endpoints that define end limits such as "no pain" and "pain as bad as possible". The patient is asked to mark the level of pain on the line between the two endpoints.

OTHER OUTCOMES:
means of blood pressure (mmHg) | up to 45 minutes
  In the study, a digital sphygmomanometer, which has been calibrated in comparison with the mercury sphygmomanometer, is used in order to prevent individual differences in the measurement of blood pressure. For accurate results, the sphygmomanometer sleeve is sized for adult individuals (width = about 20 cm, length = about 40 cm). In order for the blood pressure not to be affected by the conditions during the measurement, it is taken into account that the individual did not drink tea or coffee, take caffeine, and preferably did not eat during the 30 minutes prior to measurement.
means of heart rate (/min) | up to 45 minutes
  The heart rate is the pressure of the left ventricle on the vascular wall of the blood that it throws into the aorta during systole from the skin surface.In the research, radial heart rate is measured as manuel.
means of respiratory rate (/min) | up to 45 minutes
  The respiratory rate is the patient's breath per minute. In this study, respiratory rate was counted by monitoring chest movements for one minute while the patient was in a sitting position.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant İzzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No